CLINICAL TRIAL: NCT02957552
Title: Safety and Tolerance of Immunomodulating Therapy With Donor-specific Mesenchymal Stem Cells in Pediatric Living-Donor Liver Transplantation, a 24-month, Non-randomized, Open-label, Prospective, Single-center Pilot Trial
Brief Title: Safety and Tolerance of Immunomodulating Therapy With Donor-specific MSC in Pediatric Living-Donor Liver Transplantation
Acronym: MYSTEP1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, PD Dr. Ekkehard Sturm (MD, PhD), Head of Pediatric Gastroenterology and Hepatology, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYSTEP1; 2014-003561-15 (EudraCT Number)
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Pediatric Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with Mesenchymal Stem Cells (Experimental): Two doses of 1 x 10^6 MSCs/kg body weight:
  * first administration intraoperatively via intraportal infusion
  * second infusion via intravenous infusion on postoperative day 2 (+/- 1 day)
  Standard immunosuppressive treatment consisting of steroids, basiliximab and tacrolimus according to the center's pediatric liver transplantation protocol
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — Donor-specific, bone marrow derived mesenchymal stem (stromal) cells

SUMMARY:
Since the introduction of calcineurin-based immunosuppression, patient and graft survival in pediatric liver transplantation (LT) improved significantly. However, in contrast, calcineurin inhibitor (CNI) toxicity leads to significant morbidity and impairs quality of life for recipients. Moreover, CNI cannot prevent long-term allograft inflammation and fibrosis.

Mesenchymal stem (stromal) cells (MSC) have potent immunomodulatory properties potentially promoting allograft tolerance and ameliorating toxicity of exposure to high dose CNI. Previous trials for non-solid organ transplant indications have shown an excellent safety profile of intravenous MSC application. The MYSTEP1 trial aims to investigate safety and benefits portal and intravenous MSC infusion in pediatric LT.

DETAILED DESCRIPTION:
Background: Calcineurin inhibitors (CNI) have significantly improved patient and graft survival in pediatric liver transplantation (pLT). However, CNI toxicity leads to significant morbidity. Moreover, CNIs cannot prevent long-term allograft injury.

Mesenchymal stem (stromal) cells (MSC) have potent immunomodulatory properties, which may promote allograft tolerance and ameliorate toxicity of high-dose CNI. The MYSTEP1 trial aims to investigate safety and feasibility of donor-derived MSCs in pLT.

Methods/Design: 7 to 10 children undergoing living-donor pLT will be included in this open-label, prospective pilot trial. A dose of 1 × 106 MSCs/kg body weight will be given at two time points: first by intraportal infusion intraoperatively and second by intravenous infusion on postoperative day 2. In addition, participants will receive standard immunosuppressive treatment. Our primary objective is to assess the safety of intraportal and intravenous MSC infusion in pLT recipients. Our secondary objective is to evaluate efficacy of MSC treatment as measured by the individual need for immunosuppression and the incidence of biopsy-proven acute rejection. We will perform detailed immune monitoring to investigate immunomodulatory effects.

Discussion: Our study will provide information on the safety of donor-derived MSCs in pediatric living-donor liver transplantation and their effect on immunomodulation and graft survival.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (patients, both parents and / or legal guardian)
2. age ≥ 8 weeks and ≤ 18 years
3. undergoing living donor liver transplantation for chronic terminal liver failure
4. Body weight > 5kg

Exclusion Criteria:

1. No suitability of the living-donor
2. Pregnant or breastfeeding
3. If appropriate: no use of adequate contraception
4. Acute liver failure; highly urgent transplantations
5. Receiving any form of solid organ retransplantation
6. Multi-Organ-Transplantations
7. Active autoimmune disease
8. Pre-existing renal failure with eGFR < 50 ml/min/1.73 m2 or requiring hemodialysis
9. Reduced pulmonary function (lung function test in children older than 6 years: FEV1 and FVC < 70% of age-appropriate norm) or clinical suspicion of pulmonary disease affecting patient's physical performance, requiring invasive or non-invasive mechanical ventilation.
10. History of pulmonary embolism
11. Pulmonary hypertension and / or right ventricular load in echocardiography
12. Cardiac function: left ventricular shortening fraction (FS) < 25%
13. Clinically significant systemic infections
14. Critical care treatment like mechanical ventilation, dialysis or vasopressor agents.
15. HIV seropositive, HTLV seropositive, Hepatitis B/C seropositive
16. Hepato-biliary malignancies or history of any extra-hepatic malignancy
17. Thrombophilia
18. Budd-Chiari syndrome
19. Pre-existent thrombosis of portal vein
20. Doppler-sonographic evidence for relevant porto-systemic shunts, like persistent Ductus Venosus
21. Cold ischemia time > 90 min
22. Known abuse for drugs or alcohol
23. Known allergy to DMSO

Ages: 8 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with MYSTEP-score grade 3 and grade 2 (toxicity of MSC infusion) | 28 days
  In order to evaluate and quantifiy acute clinical complications related to MSC infusion, the investigators defined the MYSTEP score, a specific pediatric infusional toxicity scoring system (adapted from MiSOT-I score). The score focusses on description of intraportal, pulmonary and systemic toxicity. For each of these three modalities, degrees of severity between 0 (no treatment emergent adverse event) and 3 (severe treatment emergent adverse event) have been defined.
Number of participants with occurrence of any severe adverse events (SAE) | Two years
  A particular focus will be on viral infections and reactivation (ADV, HCMV, EBV, Hepatitis B, Hepatitis C and Hepatitis E), bacterial or fungal infections.
Graft function after liver transplantation - Number of participants with abnormal liver tests | Two years
  Graft function after liver transplantation, measured by aminotransferase and gamma glutamyl transferase activity, bilirubin, albumin and INR.

SECONDARY OUTCOMES:
Individual need for immunosuppressive medication | Two years
  measured by tacrolimus trough levels [ng/ml] and prednisolon dosage [mg/kgBW/day]. Tapering of tacrolimus and steroids will be performed according to a step-wise tapering protocol after day 180.
Time to first biopsy-proven acute rejection (BPAR) | Two years
  Protocol liver biopsy will be performed on day 180 post LT. Additional biopsies will be taken whenever clinically necessary.
Immune monitoring: donor-specific antibodies (DSA) | Two years
  [Participants with positive DSA]
Patient and graft survival at 1 and 2 years after liver transplantation | up to Two years
  [Death, Re-Transplantation]

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Sturm, MD, PhD, Principal Investigator — University Hospital Tuebingen, Germany; Dept. for Pediatric Gastroenterology and Hepatology
Locations (1):
- University Children's Hospital, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No